CLINICAL TRIAL: NCT07242014
Title: PET Targeting Acid Phosphatase 3 (ACP3) in Prostate Cancer and Compared With 68Ga-PSMA
Brief Title: 68Ga-XACP3 PET/CT in Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XMYY-2025KY231
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer; PET/CT; ACP3
Keywords: Prostate Cancer; PET/CT; ACP3
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-XACP3 (Experimental): Each subject receives a single intravenous injection of 68Ga-XACP3 and undergoes PET/CT imaging within the specified time.
  Interventions: Diagnostic Test: Diagnostic Test: standard-of-care imaging (68Ga-PSMA PET/CT), 68Ga-XACP3 PET/CT

INTERVENTIONS:
Diagnostic Test: Diagnostic Test: standard-of-care imaging (68Ga-PSMA PET/CT), 68Ga-XACP3 PET/CT — Each subject receives a single intravenous injection of standard-of-care imaging radiopharmaceutical (68Ga-PSMA) and 68Ga-XACP3, and undergoes PET/CT imaging within the specified time.

SUMMARY:
The objective of the study is to construct a noninvasive approach 68Ga-XACP3 PET/CT to detect tumor lesions in patients with prostate cancer and to compare with 68Ga-PSMA PET/CT.

DETAILED DESCRIPTION:
As a new ACP3 targeting PET radiotracer, 68Ga-XACP3 is promising as an excellent imaging agent applicable to prostate cancer. In this research, subjects with prostate cancer or highly suspected recurrence detection underwent contemporaneous 68Ga-XACP3 and standard-of-care imaging (68Ga-PSMA PET/CT) either for an initial assessment or for metastases or highly suspected recurrence detection. Tumor uptake was quantified by the maximum standard uptake value (SUVmax). The numbers of positive tumor lesions of standard-of-care imaging and 68Ga-PSMA PET/CT were recorded by visual interpretation. The diagnostic accuracy of 68Ga-XACP3 was calculated and compared to standard-of-care imaging.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 18 years or older);
* Patients with newly diagnosed, highly suspected recurrence or previously treated metastases of prostate cancer (supporting evidence may include MRI, CT, tumor markers, and pathology report);
* Patients who had scheduled both standard-of-care imaging (68Ga-PSMA PET/CT) and 68Ga-XACP3 PET/CT scans;
* Patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.

Exclusion Criteria:

* The inability or unwillingness of the research participant or legal representative to provide written informed consent.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic efficacy | 1 years
  Description: The sensitivity, specificity, and accuracy of standard-of-care imaging (68Ga-PSMA PET/CT) and 68Ga-XACP3 PET/CT were calculated and compared to evaluate the diagnostic accuracy.

SECONDARY OUTCOMES:
Number of lesions | 1 years
  The numbers of positive primary and metastatic lesions of standard-of-care imaging (68Ga-PSMA PET/CT) and 68Ga-XACP3 PET/CT were recorded by visual interpretation.
SUV | 1 years
  Standardized uptake value (SUV) of standard-of-care imaging (68Ga-PSMA PET/CT) and 68Ga-XACP3 PET/CT for each target lesion of subject or suspected primary tumor or/and metastasis.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No